CLINICAL TRIAL: NCT03392259
Title: Prospective Validation of Usefulness in Cardiovascular Disease (CVD) Management With CVD Management Solution Based on Interconnection to Hospital Examination
Brief Title: Usefulness of Cardiovascular Disease (CVD) Management Solution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung-Won Suh, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B-1712-438-307
Record Dates: First submitted 2018-01-01; First posted 2018-01-05 (Actual); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): conventional treatment
- App group (Experimental): conventional treatment + use of smartphone app.
  Interventions: Behavioral: Smartphone app

INTERVENTIONS:
Behavioral: Smartphone app — Installment and use of smartphone app
  Arms: App group

SUMMARY:
We previously developed the smartphone app (Heart4U) which is coupled with electronic medical record system in Seoul National University Bundang Hospital. In this study, we aim to evaluate clinical usefulness of smartphone app regarding the control of conventional risk factors in patients with history of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atherosclerotic cardiovascular diseae

  1. history of cardiovascular disease (acute myocardial infarction, unstable angina, stable angina)
  2. history of revascularization including percutaneous coronary intervention, peripheral angioplasty or bypass surgery
  3. history of stroke
  4. history of peripheral arterial disease presumed to be of atherosclerotic origin
* Patients who have smartphone and can use app by themselves
* Patients who can speak and read Korean language

Exclusion Criteria:

* Patients with evidences of delirium, confusion or impaired consciousness
* Patients who are not familiar to smartphone or app
* Patients who are not supposed to follow the study protocol adequately.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Change of 10-year ASCVD risk (10-year ASCVD risk at 6 months - 10-year ASCVD risk at baseline) | 6 months
  delta 10-year ASCVD risk between baseline and 6months, %

SECONDARY OUTCOMES:
Systolic blood pressure | 3 & 6 months
  automated blood pressure, mmHg
Diastolic blood pressure | 3 & 6 months
  automated blood pressure, mmHg
lipid profiles (total cholesterol, LDL, HDL) | 6 months
  lipid profiles at 6 months, mg/dL
body mass index | 6 months
  body mass index at 6 months, kg/m2
smoking rate | 6 months
  smoking rate at 6 months, %
degree of moderate physical activity | 6 months
  Godin Leisure-Time Exercise Questionnaire, total score (0-7)
depression scale questionnaire | 6 months
  Patient Health Questionanaire-9, total score 27 (0-27)
drug compliance | 6 months
  Medication Adherence Rating Scale (MARS), total score 10 (0-10)
App service satisfaction survey | 6 months
  Patient Activation Measure-13, total score 39 (0-39)

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Won Suh, MD, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang SH, Baek H, Cho J, Kim S, Hwang H, Lee W, Park JJ, Yoon YE, Yoon CH, Cho YS, Youn TJ, Cho GY, Chae IH, Choi DJ, Yoo S, Suh JW. Management of cardiovascular disease using an mHealth tool: a randomized clinical trial. NPJ Digit Med. 2021 Dec 3;4(1):165. doi: 10.1038/s41746-021-00535-z. PMID 34862449